CLINICAL TRIAL: NCT00416949
Title: Dose-Response in Radionuclide Therapy of Thyroid Cancer
Brief Title: Iodine I 131 in Treating Patients With Thyroid Cancer
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study was terminated due to loss of funding.
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: J0628; CDR0000522716 (Registry Identifier: PDQ (Physician Data Query)); R01CA116477-01A1 (NIH); NA_00002264 (Other: JHM IRB)
Record Dates: First submitted 2006-12-27; First posted 2006-12-28 (Estimated); Results first posted 2018-07-18 (Actual); Last update posted 2018-07-18 (Actual); Status verified 2018-06

CONDITIONS: Head and Neck Cancer
Keywords: anaplastic thyroid cancer; insular thyroid cancer; thyroid gland medullary carcinoma; recurrent thyroid cancer; stage I follicular thyroid cancer; stage I papillary thyroid cancer; stage II follicular thyroid cancer; stage II papillary thyroid cancer; stage III follicular thyroid cancer; stage III papillary thyroid cancer; stage IVA follicular thyroid cancer; stage IVB follicular thyroid cancer; stage IVC follicular thyroid cancer; stage IVA papillary thyroid cancer; stage IVB papillary thyroid cancer; stage IVC papillary thyroid cancer
MeSH Terms: conditions — Head and Neck Neoplasms; Thyroid Carcinoma, Anaplastic; Carcinoma, Medullary; Thyroid Neoplasms; Adenocarcinoma, Follicular; Thyroid Cancer, Papillary

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

ARMS (1):
- Patient-specific 3D-RD Dosimetry (Experimental): Applied a patient-specific dosimetry calculation method to the imaging data collected to calculate tumor absorbed doses, using 3D-RD method.
  Interventions: Device: Patient-specific dosimetry

INTERVENTIONS:
Device: Patient-specific dosimetry — Patient-specific 3D-RD dosimetry was applied to the data collected

SUMMARY:
RATIONALE: Radioactive iodine kills thyroid cancer cells by giving off radiation.

PURPOSE: This clinical trial is studying the side effects, best dose, and how well iodine I 131 works in treating patients with thyroid cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the relationship between estimated absorbed dose of iodine I 131 and tumor response or normal organ toxicity for different dosimetric measures, using data derived from clinical radionuclide therapy studies in patients with thyroid cancer.

OUTLINE: Patients receive oral dosimetric iodine I 131 (^131I) on day 2 and then undergo nuclear medicine imaging at 0.5-4 hours, 24, 48, and 72 hours after dosimetric ^131I. Single-photon emission computed tomography (SPECT)/CT scans are performed at 0.5-4 hours and 24 or 48 hours over the head and neck region, including the salivary glands. Subsequent SPECT/CT scans are performed over the candidate tumor sites. Patients undergo ^131I therapy on day 11.

Saliva is collected on days 1 and 2, weeks 2 and 4, and months 3 and 6 to measure saliva flow rate. Blood is collected at baseline and periodically during study to measure FLT3 ligand levels.

PROJECTED ACCRUAL: A total of 96 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of thyroid cancer
* Measurable disease by CT scan or nuclear medicine imaging
* Eligible, by standard of care criteria, for iodine I 131 therapy

PATIENT CHARACTERISTICS:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective non-barrier method contraception (e.g., combined or progesterone-only oral contraceptive pill, intrauterine device, depot progesterone, or stable relationship with a partner who has had a vasectomy)
* No other malignancy within the past 5 years except squamous cell or basal cell carcinoma of the skin
* No nonthyroidal conditions known to affect iodine I 131 uptake (e.g., New York Heart Association class III or IV congestive heart failure or renal failure)
* No alcoholism or drug abuse within the past 2 years
* No severe emotional, behavioral, or psychiatric problems that would preclude study compliance (e.g., severe claustrophobia)

PRIOR CONCURRENT THERAPY:

* No intravenous water-soluble radiographic contrast within the past 4 weeks
* No iodinated contrast agent within the past 3 months
* No concurrent drugs that may affect thyroid or renal function (e.g., renal drugs, lithium, amiodarone, other iodine-containing medication, or corticosteroids)
* No other concurrent investigational drugs

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2006-04; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: George Sgouros, PhD, Study Chair — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (1):
- Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Patient-specific 3D-RD Dosimetry
Started | 9
Completed | 4
Not Completed | 5
Not completed — Patients refused to participate | 5

BASELINE CHARACTERISTICS:
Arm/Group | Patient-specific 3D-RD Dosimetry
Number analyzed (Participants) | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 9

OUTCOME MEASURES:

1. Primary Outcome: Tumor Absorbed Dose
Description: Tumor absorbed doses (Gy) calculated using patient-specific dosimetry.
Time Frame: up to 4 years
Population: Was only able to analyze tumor data from 3 patients based on number of tumors that could be reliably imaged for analysis.
Measure: Mean (Standard Deviation); unit: Gy
Units Other Than Participants: number of tumors
Arm/Group | Patient-specific 3D-RD Dosimetry
Number analyzed (Participants) | 3
Number analyzed (number of tumors) | 5
Gy | 6.6 (4.54)

ADVERSE EVENTS:
Time Frame: 5 years
Arm/Group | Patient-specific 3D-RD Dosimetry
All-Cause Mortality (participants affected / at risk) | 0/3
Serious Adverse Events (participants affected / at risk) | 0/3
Other Adverse Events (participants affected / at risk) | 0/3

LIMITATIONS AND CAVEATS:
The protocol was designed for data collection with minimal impact on treatment. Data collection was terminated due to low accrual . No reportable results could be obtained.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No